CLINICAL TRIAL: NCT00000415
Title: Calcium Modifies Bone Response to Activity in Children
Brief Title: Physical Activity, Calcium, and Bone in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: South Dakota State University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: R01AR045310 (NIH); R01AR045310 (NIH); NIAMS-010
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Physical Activity; Nutrition
Keywords: Calcium; Physical activity; Children; Bone mass accretion; Bone mineral density (BMD); Bone response to activity and calcium supplements; Placebo; Bone growth
MeSH Terms: conditions — Motor Activity | interventions — Exercise

INTERVENTIONS:
Procedure: Physical activity
Drug: Calcium supplement

SUMMARY:
Doctors recommend that young children participate in daily physical activity to promote bone health. However, studies in adults show that physical activity and increased calcium intake cause noticeable benefits for bone health only when both factors occur together. The goal of this study is to find out whether calcium intake changes the response of bone to activity in children 3 to 4 years old. Children will participate in one of two programs conducted in childcare centers 5 days a week for 1 year. One program will involve activities that use large muscles (gross motor activity). The other will involve activities using small muscles (fine motor activity). We will give a calcium supplement (1 gram per day) to half of the children in each program and give the other half an inactive pill. We will measure bone mass and bone mineral density at the beginning and end of the study. We will take measurements 12 months after the program's completion to see if physical activity and/or calcium supplements have long-term effects on bone mineral density and physical activity.

DETAILED DESCRIPTION:
Participation in daily physical activity programs by young children is currently recommended as a means of promoting bone health. Results from studies of adults indicate that beneficial effects of either physical activity or calcium (Ca) intake may be apparent only when both these factors are present. Our results in infants indicate that physical activity combined with a low Ca diet may be detrimental in terms of bone mass accretion. The overall objective of this study is to determine whether Ca intake modifies the bone response to activity in young children 3 to 4 years of age.

Our hypotheses are that (1) the increase in bone mass resulting from a physical activity program will be more pronounced in children randomized to receive a Ca supplement compared to the increase in children randomized to receive a placebo; and (2) 12 months after cessation of the activity program, bone mass will remain higher in children randomized to gross motor activity compared to children randomized to fine motor activity, and the beneficial effect of Ca supplementation will persist only among children randomized to gross motor activity. We will test these hypotheses in a randomized 2 x 2 factorial trial in 3- to 4-year-old children. We will randomize children into either a gross motor or fine motor activity program that will be conducted in childcare centers 5 days a week for 1 year. We will further randomize each child into either a Ca supplement (1 g/d) or placebo group.

The primary outcomes of the study are bone mass accretion and changes in bone mineral density, which we will determine by dual energy x-ray absorptiometry at the beginning and end of the study. We will do activity assessments throughout the study period to determine whether participation in the gross motor activity group also increases spontaneous activity in these children. Anthropometric measurements and dietary information will allow us to statistically control for these potential confounders. We will obtain additional bone mass and physical activity measurements 12 months after completion of the program to determine if these interventions have long-term effects on bone mineral density and physical activity.

A finding of beneficial effects of Ca supplementation or physical activity, either independent of each other or in combination, will lay the groundwork for devising prevention strategies within the educational system that optimize bone health beginning early in life. However, we may find that increased physical activity in the presence of a low to moderate Ca intake may have a detrimental effect on bone mass accretion during periods of rapid growth.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in participating childcare center.
* Does not plan to attend kindergarten or withdraw from center in the next 12 months.

Exclusion Criteria:

* Chronic disease that may interfere with growth and bone mass accretion (cystic fibrosis, liver disease, asthma that is being treated with steroids, juvenile rheumatoid arthritis, immobilization).

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 224
Dates: Start 1998-04; Primary Completion 2003-02 (Actual); Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonny Specker, PhD, Principal Investigator — South Dakota State University
Locations (1):
- South Dakota State University, Brookings, South Dakota, United States

REFERENCES:
- [Background] Specker B, Binkley T. Randomized trial of physical activity and calcium supplementation on bone mineral content in 3- to 5-year-old children. J Bone Miner Res. 2003 May;18(5):885-92. doi: 10.1359/jbmr.2003.18.5.885. PMID 12733728